CLINICAL TRIAL: NCT05932992
Title: Mother Screening for Relapse Using Mid-upper Arm Circumference Among Children Recovered From Severe Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23-38829
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial of mothers being trained to measure MUAC vs standard of care to prevent relapse
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcomes assessor and investigator will be masked to intervention. In regards to the intervention, participants and care providers won't be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother screening (Active Comparator): In this arm, mothers / children dyads will be enrolled. Mothers will be trained to measure mid-upper arm circumference (MUAC) on their children weekly for 6 months. All other standard care will be provided.
  Interventions: Other: Mother education on how to perform MUAC assessment
- standard of care (No Intervention): In this arm, mothers / children dyads will be enrolled. No study intervention will be performed. all other standard of care will be provided.

INTERVENTIONS:
Other: Mother education on how to perform MUAC assessment — Mothers will be trained to perform MUAC weekly on their children
  Arms: Mother screening

SUMMARY:
The investigators propose a pilot randomized controlled trial to train mothers to screen their children post-discharge for relapse based on MUAC criteria to facilitate timely identification and referral to care for children who have relapsed.

DETAILED DESCRIPTION:
While interventions prioritizing rapid weight gain have led to improved survival for children with severe acute malnutrition (SAM), prevention of relapse to SAM after recovery is essential to improve long-term outcomes for children beyond survival. Mothers have been successfully trained to screen for new-onset SAM in community-based settings and perform as well as community health workers for detecting SAM. Here, the investigators propose a pilot randomized controlled trial in which mothers will be trained to screen their children post-discharge for relapse based on MUAC criteria to facilitate timely identification and referral to care for children who have relapsed.

SPECIFIC AIM 1: Determine the feasibility of training mothers to screen for relapse among children recovering from SAM compared to standard of care for early detection of relapse and re-entry to care. The investigators hypothesize that relapse will be detected earlier in children whose mothers have been trained to screen for relapse compared to standard of care (no mother screening).

Specific Aim 1A: Determine the burden of post-discharge relapse among children recovered from an episode of SAM in Boromo, Burkina Faso. The investigators hypothesize that >25% of children who have recovered from SAM in the study facilities will relapse within a 6-month period following their discharge.

Specific Aim 1B: Determine the acceptability and feasibility of training mothers to screen for relapse after discharge among children recovered from SAM. the investigators hypothesize that mothers will find MUAC screening acceptable and that training them will be feasible, as demonstrated by time and costs for training, willingness to participate in training, and follow-up in the trial.

SPECIFIC AIM 2: Determine the accuracy of mother-based screening for relapse among children recovering from SAM compared to a gold standard anthropometrist. the investigators hypothesize that mother screening will have a sensitivity and specificity of > 80% for the detection of relapsed SAM (MUAC < 11.5 cm) compared to screening by a trained anthropometrist.

the investigators anticipate that the result of this pilot will provide evidence supporting the acceptability, feasibility, and accuracy of mother screening for relapse among children with SAM. The data generated during this pilot will be used to support the development of a full-scale randomized controlled trial and will be used as preliminary data supporting an R01-level NIH application. These data will help establish a new line of work for our research team in the management of acute malnutrition, which builds on existing expertise in randomized controlled trials and antibiotic-based interventions for child survival and reduction of morbidity, including as part of the management of uncomplicated SAM.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver's aged 18 years old or older or a legal guardian or a relative aged 18 or older
* Child aged 6-59 months
* Child has recovered from an episode of SAM per Burkinabè national guidelines (WHZ ≥

  * 2 and/or MUAC ≥ 12.5 cm in the past month
* Family is planning to stay in the study area for 6 months
* Appropriate consent from the caregiver or guardian

Exclusion Criteria:

* Caregiver age under 18 years old, or legal guardian or relatives under 18 years old
* Child age < 6 months or > 59 months
* Twins/multiple births and children with feeding issues
* Did not recover from SAM in the past month
* Family is planning to move out of the study area in the next 6 months
* Caregiver or guardian refuses to provide consent

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Time to detection of relapse | 6 months
  Time to relapse using a log-rank test with a term for randomized treatment assignment will be used.
  Relapse will be defined using the Burkina Faso guideline for detecting malnutrition (MUAC < 11.5 cm and / or weight-for-height Z-scores WHZ < -3 SD)

SECONDARY OUTCOMES:
Weight for Height Z score (WHZ) | 6 months
  Weight for Height Z score will be calculated and compared between arms
weight-for-age Z-score (WAZ) | 6 months
  weight-for-age Z-score will be calculated and compared between arms
height-for-age Z-score (HAZ) | 6 months
  height-for-age Z-score will be calculated and compared between arms

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Oldenburg, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- Centre de recherche en sante de nouna, Nouna, Burkina Faso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bountogo M, Dah C, Ouedraogo M, Zerbo F, Kouanda I, Lebas E, Fetterman I, La Mons J, Burroughs H, Arnold BF, Sie A, Oldenburg CE. Caregiver Screening for Relapse Among Children Recently Recovered From Severe Acute Malnutrition: A Randomized Controlled Feasibility Trial. Matern Child Nutr. 2026 Mar;22(1):e70160. doi: 10.1111/mcn.70160. PMID 41569394
- [Derived] Dah C, Kimfuema A, Bountogo M, Zerbo F, Ouedraogo M, Kouanda I, Fetterman I, Arnold BF, Lebas E, Sie A, Oldenburg CE. Training caregivers to screen for relapse among children who have recovered from severe acute malnutrition: study protocol for a feasibility trial. Pilot Feasibility Stud. 2026 Jan 13. doi: 10.1186/s40814-025-01752-z. Online ahead of print. PMID 41527000